CLINICAL TRIAL: NCT07275892
Title: Pilot Feasibility Trial of a Peer Support Program for Trauma Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marina Wasilewski, Senior Scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 6905
Record Dates: First submitted 2025-09-04; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Injury; Burns; Amputation; Mental Health Outcomes
Keywords: Peer Support; Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Intervention Model Description: Trauma survivors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm pilot feasibility study (Experimental): To evaluate implementation and preliminary impact prior to a future RCT.
  Interventions: Behavioral: Cross-continuum Peer Support Program

INTERVENTIONS:
Behavioral: Cross-continuum Peer Support Program — Trained trauma-survivor peer supporters (n=4), supported by a research team member; peers complete a 5-session training covering trauma-informed communication, boundaries, crisis de-escalation, self-care, and secondary trauma. Trauma survivors will be recruited in acute care and have the option to meeting once with a trained peer supporter prior to discharge to inpatient rehabilitation. In in-patient rehab they will attend 1 hour peer support group sessions facilitated by the trained peer supporters twice a week for a total of 3 weeks. Once discharged the community, they will attend 1 hour peer support group sessions facilitated by the trained peer supporters once a week for a total of 12 weeks.

SUMMARY:
Traumatic injuries from events like car crashes, falls, or fires are a leading cause of disability. Survivors often face not only physical challenges but also long-lasting pain, mental health challenges and difficulty returning to work and family life. Although medical care focuses on physical recovery, survivors frequently report that their emotional and social needs are overlooked and unmet.

Peer support-guidance from people who have lived through similar injuries-can reduce distress and improve coping. However, no programs in Canada currently provide peer support to trauma survivors across their recovery journey, from hospital to rehabilitation to community living.

The investigators worked with trauma survivors, caregivers, and healthcare providers to co-design a Peer Support Program (PSP) that offers support throughout these stages. This pilot study will test whether the program is feasible and acceptable, and explore its early impact on recovery. Results will guide a future larger trial to expand peer support in trauma care.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years+) who have experienced an unintentional traumatic injury resulting in hospitalization at Sunnybrook and who will be discharged to inpatient rehabilitation at St. John's Rehab after acute care.
* must be able to communicate in English

Exclusion Criteria:

* patients who experienced: a) an intentional self-harm injury (because self-harm suggests a history of mental health issues prior to the trauma requiring specific psychiatric supports)
* patients who experienced: an injury caused by an intimate partner (because these injuries are typically underpinned by chronic exposure to domestic violence which requires interventions that promote patient safety and interrupt the pattern of violence)
* patients who experienced: a violently-acquired injury (as this patient population already receives specific clinical and social support through Sunnybrook's BReAking the Cycle of Violence with Empathy (BRAVE) program).
* patients with substantial cognitive impairment and a history of substance misuse if their HCPs indicate that either condition will impede the their ability to provide informed consent and/or participate safely in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the Peer Support Program | From recruitment to 3 months post intervention
  To determine the feasibility of implementing the Peer Support Program (PSP) for trauma survivors. We will measure the criteria below to establish feasibility. These feasibility goals were established with reference to another study our group conducted aimed at assessing the feasibility of a novel psychosocial group intervention for amputees.
  * RECRUITMENT (proportion of eligible participants approached who consent-GOAL: ≥50%),
  * WITHDRAWAL (proportion of study participants who withdraw from the study before the end of Phase II (Inpatient Rehabilitation)-GOAL: ≤ 25%)
  * ADHERENCE (proportion of PSP sessions attended by participants-GOAL: ≥60%),
  * RETENTION (proportion of participants who complete the program-GOAL: ≥60%);
  * BASELINE SURVEYS (proportion of surveys completed-GOAL: ≥70%).
  * POST-INTERVENTION SURVEY (proportion of surveys completed-GOAL: ≥60%):
  * SURVEY AT 3 MONTH FOLLOW UP (proportion of surveys completed-GOAL: ≥50%):

SECONDARY OUTCOMES:
Community Reintegration - Normal Living Index (RNL) Index | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The 11-item Reintegration to Normal Living Index (RNL) Index covers areas such as involvement in recreational and social activities, perceived ability to move within the community, and the degree of comfort people have with their relationships. It is a valid and reliable tool for assessing participation in various populations. Scores range from 0 to 110, with a higher score indicating a higher level of community reintegration.
Coping Self-Efficacy (CSE) - 20-item CSE Scale | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The 20-item CSE Scale66 is a coping self-efficacy scale that has a robust factor structure across different types of post-traumatic events, making it especially suitable for use in various trauma populations. For each item, respondents rate their perceived efficacy on dealing with different consequences of trauma on a 7-point scale (e.g. 'resuming normal life'; 'being optimistic since the event'). Scores range from 20 (low self-efficacy) to 140 (high self-efficacy). The internal consistency of the scale has been found to be excellent across three panel waves of data in persons who had experienced a traumatic event in the previous two years
Health-Related Quality of Life - The Short-Form 36 (SF-36) | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The Short-Form 36 (SF-36) is the most widely used generic health-related QoL instrument, including Neuro-musculoskeletal injuries, which measures 8 multi-item dimensions of health: physical functioning, social functioning, role limitations due to physical and emotional problems, mental health, energy/vitality, pain, and general health perception. Scores range from 0 to 100 on each domain, with lower scores indicating poorer function. These eight dimensions are summarized into a physical and mental health summary score. The SF-36 is sensitive to changes in functioning over time, and has demonstrated clinically meaningful, albeit modest, change in trauma patients.
Post-Traumatic Stress Disorder (PTSD) - The PTSD Checklist-Civilian Version (PCL-C) | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The PTSD Checklist-Civilian Version (PCL-C) is a standardized 17-item self-report rating scale for PTSD that is well-validated across different populations. Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point scale, with higher scores indicating more severe levels of PTSD.
Post-Traumatic Growth - The Post-Traumatic Growth Inventory (PTGI) | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The Post-Traumatic Growth Inventory (PTGI) is a 21-item scale assessing positive outcomes reported by those who have experienced traumatic events. Items are scored on a 6-point scale and scores range from 0 to 105, with higher scores indicating greater levels of growth. It has good levels of internal consistency reliability (α=.90) and 2-month test-retest stability (r =.71).
Social Support - The Medical Outcomes Study Social Support Survey (MOS-SS) | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The Medical Outcomes Study Social Support Survey (MOS-SS) is a 19-item measure of perceived social support across four subscales: emotional/information support; tangible support; affectionate support; and positive social interaction. Questions are answered on a 5-point scale ranging from "none of the time" to "all of the time", with higher scores indicating more support. The MOS-SS has very good internal consistency across populations including chronic disease and chronic pain.
Loneliness and Social Isolation -The UCLA 3-Item Loneliness Scale | Baseline, up to 2 weeks post intervention, and 3-months post intervention
  The UCLA 3-Item Loneliness Scale measures three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. Items are scored from 1 (hardly ever) to 3 (often), with higher scores indicating greater loneliness and isolation. It has satisfactory reliability and both concurrent and discriminant validity.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Wasilewski, PhD, Principal Investigator — St. John's Rehab Research Program, Sunnybrook Research Institute, Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - St. John's Rehab at Sunnybrook, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
To maintain patient confidentiality.

REFERENCES:
- [Background] Dennis CL. Peer support within a health care context: a concept analysis. Int J Nurs Stud. 2003 Mar;40(3):321-32. doi: 10.1016/s0020-7489(02)00092-5. PMID 12605954
- [Background] Braun V, Clarke V. Reflecting on reflexive thematic analysis. Qualitative research in sport, exercise and health. 2019;11(4):589-597
- [Background] Braun V, Clarke V. One size fits all? What counts as quality practice in (reflexive) thematic analysis? Qualitative research in psychology. 2021;18(3):328-352
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology. 2006/01/01 2006;3(2):77-101. doi:10.1191/1478088706qp063oa
- [Background] Hitzig SL, Gotlib Conn L, Guilcher SJT, Cimino SR, Robinson LR. Understanding the role of the physiatrist and how to improve the continuum of care for trauma patients: a qualitative study. Disabil Rehabil. 2021 Oct;43(20):2846-2853. doi: 10.1080/09638288.2020.1719215. Epub 2020 Feb 4. PMID 32017865
- [Background] Wasilewski MB, Stinson JN, Webster F, Cameron JI. Using Twitter to recruit participants for health research: An example from a caregiving study. Health Informatics J. 2019 Dec;25(4):1485-1497. doi: 10.1177/1460458218775158. Epub 2018 May 30. PMID 29843545
- [Background] Thorogood N, Green J. Qualitative Methods for Health Research. SAGE Publications Ltd.; 2009
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Ljungvall H, Ekselius L, Asenlof P. Reliability, construct validity, and factorial structure of a Swedish version of the medical outcomes study social support survey (MOS-SSS) in patients with chronic pain. Scand J Pain. 2023 Sep 18;24(1). doi: 10.1515/sjpain-2023-0002. eCollection 2024 Jan 1. PMID 37712773
- [Background] Merino-Soto C, Nunez Benitez MA, Dominguez-Guedea MT, Toledano-Toledano F, Moral de la Rubia J, Astudillo-Garcia CI, Rivera-Rivera L, Leyva-Lopez A, Angulo-Ramos M, Flores Laguna OA, Hernandez-Salinas G, Rodriguez Castro JH, Gonzalez Pena OI, Garduno Espinosa J. Medical outcomes study social support survey (MOS-SSS) in patients with chronic disease: A psychometric assessment. Front Psychiatry. 2023 Jan 11;13:1028342. doi: 10.3389/fpsyt.2022.1028342. eCollection 2022. PMID 36713918
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Wilkins KC, Lang AJ, Norman SB. Synthesis of the psychometric properties of the PTSD checklist (PCL) military, civilian, and specific versions. Depress Anxiety. 2011 Jul;28(7):596-606. doi: 10.1002/da.20837. Epub 2011 Jun 16. PMID 21681864
- [Background] Pan SL, Liang HW, Hou WH, Yeh TS. Responsiveness of SF-36 and Lower Extremity Functional Scale for assessing outcomes in traumatic injuries of lower extremities. Injury. 2014 Nov;45(11):1759-63. doi: 10.1016/j.injury.2014.05.022. Epub 2014 May 28. PMID 24938677
- [Background] Kaske S, Lefering R, Trentzsch H, Driessen A, Bouillon B, Maegele M, Probst C. Quality of life two years after severe trauma: a single-centre evaluation. Injury. 2014 Oct;45 Suppl 3:S100-5. doi: 10.1016/j.injury.2014.08.028. PMID 25284226
- [Background] Mackenzie EJ, Rivara FP, Jurkovich GJ, Nathens AB, Egleston BL, Salkever DS, Frey KP, Scharfstein DO. The impact of trauma-center care on functional outcomes following major lower-limb trauma. J Bone Joint Surg Am. 2008 Jan;90(1):101-9. doi: 10.2106/JBJS.F.01225. PMID 18171963
- [Background] Gopinath B, Harris IA, Nicholas M, Casey P, Blyth F, Maher CG, Cameron ID. A comparison of health outcomes in older versus younger adults following a road traffic crash injury: a cohort study. PLoS One. 2015 Apr 1;10(4):e0122732. doi: 10.1371/journal.pone.0122732. eCollection 2015. PMID 25830702
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Benight CC, Shoji K, James LE, Waldrep EE, Delahanty DL, Cieslak R. Trauma Coping Self-Efficacy: A Context-Specific Self-Efficacy Measure for Traumatic Stress. Psychol Trauma. 2015 Nov;7(6):591-599. doi: 10.1037/tra0000045. PMID 26524542
- [Background] Bosmans MW, van der Velden PG. Longitudinal interplay between posttraumatic stress symptoms and coping self-efficacy: A four-wave prospective study. Soc Sci Med. 2015 Jun;134:23-9. doi: 10.1016/j.socscimed.2015.04.007. Epub 2015 Apr 9. PMID 25875423
- [Background] Udayar S, Urbanaviciute I, Rossier J. Perceived social support and Big Five personality traits in middle adulthood: A 4-year cross-lagged path analysis. Applied Research in Quality of Life. 2020;15:395-414
- [Background] Polman R, Borkoles E, Nicholls AR. Type D personality, stress, and symptoms of burnout: the influence of avoidance coping and social support. Br J Health Psychol. 2010 Sep;15(Pt 3):681-96. doi: 10.1348/135910709X479069. Epub 2009 Nov 21. PMID 19930789
- [Background] Jaksic N, Brajkovic L, Ivezic E, Topic R, Jakovljevic M. The role of personality traits in posttraumatic stress disorder (PTSD). Psychiatr Danub. 2012 Sep;24(3):256-66. PMID 23013628
- [Background] Gosling SD, Rentfrow PJ, Swann Jr WB. A very brief measure of the Big-Five personality domains. Journal of Research in personality. 2003;37(6):504-528
- [Background] Holzer LA, Sevelda F, Fraberger G, Bluder O, Kickinger W, Holzer G. Body image and self-esteem in lower-limb amputees. PLoS One. 2014 Mar 24;9(3):e92943. doi: 10.1371/journal.pone.0092943. eCollection 2014. PMID 24663958
- [Background] Singh R, Hunter J, Philip A, Tyson S. Gender differences in amputation outcome. Disabil Rehabil. 2008;30(2):122-5. doi: 10.1080/09638280701254095. PMID 17852206
- [Background] Holbrook TL, Hoyt DB, Stein MB, Sieber WJ. Gender differences in long-term posttraumatic stress disorder outcomes after major trauma: women are at higher risk of adverse outcomes than men. J Trauma. 2002 Nov;53(5):882-8. doi: 10.1097/00005373-200211000-00012. PMID 12435938
- [Background] Holbrook TL, Hoyt DB, Anderson JP. The importance of gender on outcome after major trauma: functional and psychologic outcomes in women versus men. J Trauma. 2001 Feb;50(2):270-3. doi: 10.1097/00005373-200102000-00012. PMID 11242291
- [Background] McCarthy ML, MacKenzie EJ, Bosse MJ, Copeland CE, Hash CS, Burgess AR. Functional status following orthopedic trauma in young women. J Trauma. 1995 Nov;39(5):828-36; discussion 836-7. doi: 10.1097/00005373-199511000-00005. PMID 7473997
- [Background] Santiago PN, Ursano RJ, Gray CL, Pynoos RS, Spiegel D, Lewis-Fernandez R, Friedman MJ, Fullerton CS. A systematic review of PTSD prevalence and trajectories in DSM-5 defined trauma exposed populations: intentional and non-intentional traumatic events. PLoS One. 2013 Apr 11;8(4):e59236. doi: 10.1371/journal.pone.0059236. Print 2013. PMID 23593134
- [Background] Jiang T, Webster JL, Robinson A, Kassam-Adams N, Richmond TS. Emotional responses to unintentional and intentional traumatic injuries among urban black men: A qualitative study. Injury. 2018 May;49(5):983-989. doi: 10.1016/j.injury.2017.12.002. Epub 2017 Dec 6. PMID 29248186
- [Background] Nicholls SG, Fox G, Monfaredi Z, Poole E, Garritty C, Maybee A, Presseau J, Shea B, Fergusson DA. The impact of patient engagement on trials and trialists in Ontario, Canada: An interview study with IMPACT awardees. Res Involv Engagem. 2022 Sep 7;8(1):50. doi: 10.1186/s40900-022-00381-7. PMID 36071496
- [Background] Kynoch K, Ramis MA. Experience based co-design in acute healthcare services: a scoping review protocol. JBI Database System Rev Implement Rep. 2019 Jan;17(1):3-9. doi: 10.11124/JBISRIR-2017-003655. PMID 30024434
- [Background] Straus SE, Tetroe J, Graham ID. Knowledge translation in health care: moving from evidence to practice. John Wiley & Sons; 2013
- [Background] Shahsavari H, Matourypour P, Ghiyasvandian S, Nejad MRG. Medical Research Council framework for development and evaluation of complex interventions: A comprehensive guidance. J Educ Health Promot. 2020 Apr 28;9:88. doi: 10.4103/jehp.jehp_649_19. eCollection 2020. No abstract available. PMID 32509896
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Magasi S, Papadimitriou C. Peer Support Interventions in Physical Medicine and Rehabilitation: A Framework to Advance the Field. Arch Phys Med Rehabil. 2022 Jul;103(7S):S222-S229. doi: 10.1016/j.apmr.2020.09.400. Epub 2021 Jan 10. PMID 33440133
- [Background] Hope V. Understanding the Cost Effectiveness of Using Peer Specialists From : Via Hope. (2012). Peer Specialist Integration Workbook. Austin, Texas: Via Hope. 2012. http://sites.utexas.edu/mental-health-institute/files/2012/10/Understanding_the_Cost_Effectiveness_of_Using_Peer_Specialists.pdf
- [Background] American Trauma Society. Trauma Suvivors Network. Accessed 1/29/2020, 2020. www.traumasurvivorsnetwork.org
- [Background] Haines KJ, Beesley SJ, Hopkins RO, McPeake J, Quasim T, Ritchie K, Iwashyna TJ. Peer Support in Critical Care: A Systematic Review. Crit Care Med. 2018 Sep;46(9):1522-1531. doi: 10.1097/CCM.0000000000003293. PMID 29957717
- [Background] Hanks RA, Rapport LJ, Wertheimer J, Koviak C. Randomized controlled trial of peer mentoring for individuals with traumatic brain injury and their significant others. Arch Phys Med Rehabil. 2012 Aug;93(8):1297-304. doi: 10.1016/j.apmr.2012.04.027. PMID 22840826
- [Background] Gassaway J, Jones ML, Sweatman WM, Hong M, Anziano P, DeVault K. Effects of Peer Mentoring on Self-Efficacy and Hospital Readmission After Inpatient Rehabilitation of Individuals With Spinal Cord Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1526-1534.e2. doi: 10.1016/j.apmr.2017.02.018. Epub 2017 Mar 23. PMID 28342829
- [Background] Institute of Medicine (US) Committee on Injury Prevention and Control; Bonnie RJ, Fulco CE, Liverman CT, editors. Reducing the Burden of Injury: Advancing Prevention and Treatment. Washington (DC): National Academies Press (US); 1999. Available from http://www.ncbi.nlm.nih.gov/books/NBK230590/ PMID 25101422
- [Background] Virani T. Development of a Peer Support Strategy for the South West LHIN. 2015
- [Background] Progress Pf. Economic Analysis of Peer Support Programs. 2015. http://peersforprogress.org/wp-content/uploads/2015/04/150417-economic-analysis-in-peer-support.pdf
- [Background] House JS. Work stress and social support. Addison-Wesley series on occupational stress ; 4. Addison-Wesley Pub. Co; 1981
- [Background] Mental Health Foundation. Peer support. Accessed 12/17/2019, https://www.mentalhealth.org.uk/a-to-z/p/peer-support
- [Background] Reichmann JP, Bartman KR. An integrative review of peer support for patients undergoing major limb amputation. J Vasc Nurs. 2018 Mar;36(1):34-39. doi: 10.1016/j.jvn.2017.10.002. Epub 2017 Nov 22. PMID 29452628
- [Background] Waites B, Zigmond A. Psychological impact of amputation. Therapy for Amputees 3rd ed Edinburg: Churchill Livingstone. 1999:27-39
- [Background] Mental Health Foundation. Peer Support. Accessed 01/08/2020, https://www.mentalhealth.org.uk/a-to-z/p/peer-support
- [Background] Jones M, Gassaway J. Peer-supported self-management to facilitate community re-entry after discharge from spinal cord injury rehabilitation: Engaging peers as change agents and research partners. Annals of physical and rehabilitation medicine. 2016;59:e128-e129
- [Background] Zatzick D, Russo J, Thomas P, Darnell D, Teter H, Ingraham L, Whiteside LK, Wang J, Guiney R, Parker L, Sandgren K, Hedrick MK, Van Eaton EG, Jurkovich G. Patient-Centered Care Transitions After Injury Hospitalization: A Comparative Effectiveness Trial. Psychiatry. 2018 Summer;81(2):141-157. doi: 10.1080/00332747.2017.1354621. Epub 2018 Mar 13. PMID 29533154
- [Background] Hibbard MR, Cantor J, Charatz H, Rosenthal R, Ashman T, Gundersen N, Ireland-Knight L, Gordon W, Avner J, Gartner A. Peer support in the community: initial findings of a mentoring program for individuals with traumatic brain injury and their families. J Head Trauma Rehabil. 2002 Apr;17(2):112-31. doi: 10.1097/00001199-200204000-00004. PMID 11909510
- [Background] Haas B, Jeon SH, Rotermann M, Stepner M, Fransoo R, Sanmartin C, Wunsch H, Scales DC, Iwashyna TJ, Garland A. Association of Severe Trauma With Work and Earnings in a National Cohort in Canada. JAMA Surg. 2021 Jan 1;156(1):51-59. doi: 10.1001/jamasurg.2020.4599. PMID 33112383
- [Background] Blakeney PE, Rosenberg L, Rosenberg M, Faber AW. Psychosocial care of persons with severe burns. Burns. 2008 Jun;34(4):433-40. doi: 10.1016/j.burns.2007.08.008. Epub 2008 Jan 18. PMID 18207643
- [Background] Ponzer S, Molin U, Johansson SE, Bergman B, Tornkvist H. Psychosocial support in rehabilitation after orthopedic injuries. J Trauma. 2000 Feb;48(2):273-9. doi: 10.1097/00005373-200002000-00013. PMID 10697086
- [Background] Sullivan MJ, Ward LC, Tripp D, French DJ, Adams H, Stanish WD. Secondary prevention of work disability: community-based psychosocial intervention for musculoskeletal disorders. J Occup Rehabil. 2005 Sep;15(3):377-92. doi: 10.1007/s10926-005-5944-7. PMID 16119228
- [Background] Lee KH, Chua J. Psychosocial Support Following Maxillofacial Trauma and its Impact on Trauma Recurrence. J Maxillofac Oral Surg. 2018 Mar;17(1):32-37. doi: 10.1007/s12663-016-0979-2. Epub 2016 Oct 18. PMID 29382991
- [Background] Zatzick DF, Roy-Byrne P, Russo JE, Rivara FP, Koike A, Jurkovich GJ, Katon W. Collaborative interventions for physically injured trauma survivors: a pilot randomized effectiveness trial. Gen Hosp Psychiatry. 2001 May-Jun;23(3):114-23. doi: 10.1016/s0163-8343(01)00140-2. PMID 11427243
- [Background] Major Extremity Trauma Rehabilitation Consortium (METRC). Early Effects of the Trauma Collaborative Care Intervention: Results From a Prospective Multicenter Cluster Clinical Trial. J Orthop Trauma. 2019 Nov;33(11):538-546. doi: 10.1097/BOT.0000000000001581. PMID 31634286
- [Background] De Silva M, Maclachlan M, Devane D, Desmond D, Gallagher P, Schnyder U, Brennan M, Patel V. Psychosocial interventions for the prevention of disability following traumatic physical injury. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD006422. doi: 10.1002/14651858.CD006422.pub3. PMID 19821365
- [Background] Shalev AY, Ankri Y, Israeli-Shalev Y, Peleg T, Adessky R, Freedman S. Prevention of posttraumatic stress disorder by early treatment: results from the Jerusalem Trauma Outreach And Prevention study. Arch Gen Psychiatry. 2012 Feb;69(2):166-76. doi: 10.1001/archgenpsychiatry.2011.127. Epub 2011 Oct 3. PMID 21969418
- [Background] Petrie M, Zatzick D. Collaborative care interventions in general trauma patients. Oral Maxillofac Surg Clin North Am. 2010 May;22(2):261-7. doi: 10.1016/j.coms.2010.01.002. PMID 20403558
- [Background] Bosse MJ, MacKenzie EJ, Kellam JF, Burgess AR, Webb LX, Swiontkowski MF, Sanders RW, Jones AL, McAndrew MP, Patterson BM, McCarthy ML, Travison TG, Castillo RC. An analysis of outcomes of reconstruction or amputation after leg-threatening injuries. N Engl J Med. 2002 Dec 12;347(24):1924-31. doi: 10.1056/NEJMoa012604. PMID 12477942
- [Background] Hitzig S, Babatunde F, Colantonio A, et al. Developing a Patient-Oriented Rehabilitation Research Agenda. Toronto, ON, Canada: CIHR; 2018
- [Background] Gotlib Conn L, Zwaiman A, DasGupta T, Hales B, Watamaniuk A, Nathens AB. Trauma patient discharge and care transition experiences: Identifying opportunities for quality improvement in trauma centres. Injury. 2018 Jan;49(1):97-103. doi: 10.1016/j.injury.2017.09.028. Epub 2017 Sep 28. PMID 28988066
- [Background] Bradford AN, Castillo RC, Carlini AR, Wegener ST, Teter H Jr, Mackenzie EJ. The trauma survivors network: Survive. Connect. Rebuild. J Trauma. 2011 Jun;70(6):1557-60. doi: 10.1097/TA.0b013e3182196e7e. PMID 21817993
- [Background] Danielsson FB, Schultz Larsen M, Norgaard B, Lauritsen JM. Quality of life and level of post-traumatic stress disorder among trauma patients: A comparative study between a regional and a university hospital. Scand J Trauma Resusc Emerg Med. 2018 Jun 1;26(1):44. doi: 10.1186/s13049-018-0507-0. PMID 29859111
- [Background] Evans CCD, DeWit Y, Seitz D, Mason S, Nathens A, Hall S. Mental health outcomes after major trauma in Ontario: a population-based analysis. CMAJ. 2018 Nov 12;190(45):E1319-E1327. doi: 10.1503/cmaj.180368. PMID 30420387
- [Background] Vincent HK, Horodyski M, Vincent KR, Brisbane ST, Sadasivan KK. Psychological Distress After Orthopedic Trauma: Prevalence in Patients and Implications for Rehabilitation. PM R. 2015 Sep;7(9):978-989. doi: 10.1016/j.pmrj.2015.03.007. Epub 2015 Mar 12. PMID 25772720
- [Background] Peterson C, Miller GF, Barnett SBL, Florence C. Economic Cost of Injury - United States, 2019. MMWR Morb Mortal Wkly Rep. 2021 Dec 3;70(48):1655-1659. doi: 10.15585/mmwr.mm7048a1. PMID 34855726
- [Background] Pope AM, Tarlov AR. Disability in America: Toward a national agenda for prevention. ERIC; 1991
- [Background] Castillo RC, Raja SN, Frey KP, Vallier HA, Tornetta P 3rd, Jaeblon T, Goff BJ, Gottschalk A, Scharfstein DO, O'Toole RV; METRC. Improving Pain Management and Long-Term Outcomes Following High-Energy Orthopaedic Trauma (Pain Study). J Orthop Trauma. 2017 Apr;31 Suppl 1:S71-S77. doi: 10.1097/BOT.0000000000000793. PMID 28323806
- [Background] Lambers K, Ootes D, Ring D. Incidence of patients with lower extremity injuries presenting to US emergency departments by anatomic region, disease category, and age. Clin Orthop Relat Res. 2012 Jan;470(1):284-90. doi: 10.1007/s11999-011-1982-z. Epub 2011 Jul 22. PMID 21785896
- [Background] Nawar EW, Niska RW, Xu J. National Hospital Ambulatory Medical Care Survey: 2005 emergency department summary. Adv Data. 2007 Jun 29;(386):1-32. PMID 17703794
- [Background] Levitt EB, Patch DA, Hess MC, Terrero A, Jaeger B, Haendel MA, Chute CG, Yeager MT, Ponce BA, Theiss SM, Spitler CA, Johnson JP. Outcomes of SARS-CoV-2 infection among patients with orthopaedic fracture surgery in the National COVID Cohort Collaborative (N3C). Injury. 2023 Dec;54(12):111092. doi: 10.1016/j.injury.2023.111092. Epub 2023 Oct 12. PMID 37871347
- [Background] Organization WH. The global burden of disease: 2004 update. World Health Organization; 2008
- [Background] Haagsma JA, Graetz N, Bolliger I, Naghavi M, Higashi H, Mullany EC, Abera SF, Abraham JP, Adofo K, Alsharif U, Ameh EA, Ammar W, Antonio CA, Barrero LH, Bekele T, Bose D, Brazinova A, Catala-Lopez F, Dandona L, Dandona R, Dargan PI, De Leo D, Degenhardt L, Derrett S, Dharmaratne SD, Driscoll TR, Duan L, Petrovich Ermakov S, Farzadfar F, Feigin VL, Franklin RC, Gabbe B, Gosselin RA, Hafezi-Nejad N, Hamadeh RR, Hijar M, Hu G, Jayaraman SP, Jiang G, Khader YS, Khan EA, Krishnaswami S, Kulkarni C, Lecky FE, Leung R, Lunevicius R, Lyons RA, Majdan M, Mason-Jones AJ, Matzopoulos R, Meaney PA, Mekonnen W, Miller TR, Mock CN, Norman RE, Orozco R, Polinder S, Pourmalek F, Rahimi-Movaghar V, Refaat A, Rojas-Rueda D, Roy N, Schwebel DC, Shaheen A, Shahraz S, Skirbekk V, Soreide K, Soshnikov S, Stein DJ, Sykes BL, Tabb KM, Temesgen AM, Tenkorang EY, Theadom AM, Tran BX, Vasankari TJ, Vavilala MS, Vlassov VV, Woldeyohannes SM, Yip P, Yonemoto N, Younis MZ, Yu C, Murray CJ, Vos T. The global burden of injury: incidence, mortality, disability-adjusted life years and time trends from the Global Burden of Disease study 2013. Inj Prev. 2016 Feb;22(1):3-18. doi: 10.1136/injuryprev-2015-041616. Epub 2015 Dec 3. PMID 26635210